CLINICAL TRIAL: NCT01792635
Title: A 6-week Phase 2a Randomized, Double-blind, Placebo-controlled, Parallel Group Study To Assess Safety, Tolerability And Pharmacodynamics Of Oral Pf-05175157 As Monotherapy In Subjects With Type 2 Diabetes Mellitus
Brief Title: A 6-Week Study Of PF-05175157 In Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely on 16 May 2014 due to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731003
Record Dates: First submitted 2012-12-20; First posted 2013-02-15 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Pharmacodynamics; Safety & Tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Pilot Study) (No Intervention)
- Monotherapy (Part B) (Experimental)
  Interventions: Drug: PF-05175157; Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — PF-05175157 will be administered at 200 mg twice a day for 43 days.
  Arms: Monotherapy (Part B)
Drug: Placebo — Placebo tablets matched to PF-05175157 will be administered twice a day for 43 days.
  Arms: Monotherapy (Part B)

SUMMARY:
This study is designed to assess the safety, tolerability and pharmacodynamics of 6 weeks of oral doses of PF-05175157 provided as monotherapy in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been diagnosed with type 2 diabetes mellitus by a medical professional according to the American Diabetes Association guidelines.
* Hemoglobin A1c of ≥7 and ≤10.0% in subjects who are metformin-naive or have not taken metformin for 2 months or Hemoglobin A1c of ≥6.5 and ≤9.5% in subjects who are metformin-naïve and are taking SU or DPP-IVi which is washed off or taking metformin and are willing to discontinue metformin in a 8-week washout period.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine (other than T2DM and hypothyroidism), gastrointestinal, cardiovascular, pulmonary, hepatic, psychiatric or neurologic disease.
* A waist circumference which makes fitting imto the bore of the MR scanner impossible.

Subjects with history of dry eye, known ocular or systemic disease that affect the sclera or cornea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731003&StudyName=A%206-Week%20Study%20Of%20PF-05175157%20In%20Type%202%20Diabetes%20Mellitus

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants in Part A: Participants underwent 2 step euglycemic hyperinsulinemic clamp procedure and were infused with insulin according to a specified algorithm to reduce plasma glucose levels to approximately 100 milligram (mg)/deciliter (dL). In Step 1 of the clamp, each individual's insulin infusion rate during the last 2 hours of the overnight infusion was increased by 10 mU/square meter (m^2)/minute (min). During Step 2, all participants received an insulin infusion, at a rate of 120 mU/m^2/min.
- Placebo - Part B: Participants received placebo twice a day at approximately 08:00 immediately before the morning meal, and at approximately 18:00 before the dinner meal. The treatment period was 6 weeks.
- PF-05175157 200 mg Twice a Day - Part B: Participants received PF-05175157 200 mg twice a day at approximately 08:00 immediately before the morning meal, and at approximately 18:00 before the dinner meal. The treatment period was 6 weeks.
Period: Part A
Arm/Group | All Participants in Part A | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B
Arm/Group | All Participants in Part A | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Started | 0 | 6 | 7
Completed | 0 | 2 | 3
Not Completed | 0 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Study terminated | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All Participants in Part A | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B | Total
Number analyzed (Participants) | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.7 (9.5) | 49.3 (9.2) | 55.1 (4.6) | 51.9 (7.9)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 5 | 5 | 5 | 15
  Female | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Glucose Infusion Rates (GIR) in Part A
Description: GIR obtained averaging respectively the last 30 minutes of glucose infusion at steady state on Step 1 (ie 150 to 180 min) and Step 2 (ie 330 to 360 min) insulin infusion. Whole-body insulin sensitivity was assessed with the euglycemic hyperinsulinemic clamp procedure; the use of 2 stepped insulin infusions and labeled glucose allowed the differentiation between hepatic and peripheral insulin sensitivity. Assessment of whole body insulin sensitivity was performed during the steady states of the low insulin infusion rate (ie, Step 1) and during the steady state of the high insulin infusion rate (ie, Step 2). These indices were called GIR1 and GIR2, respectively.
Time Frame: 1 day
Population: All participants randomized and who had at least one euglycemic hyperinsulinemic clamp
Measure: Mean (90% Confidence Interval); unit: mg/min
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
mg/min
  Clamp 1 GIR1 | 191 [153 to 229]
  Clamp 1 GIR2 | 780 [580 to 980]
  Clamp 2 GIR1 | 152 [132 to 172]

2. Primary Outcome: Endogenous Gucose Production (EGP) in Part A
Description: EGP measured by means of euglycemic hyperinsulinemic clamp preceding insulin infusion (EGP0), on Step 1 insulin infusion (EGP1) and on Step 2 insulin infusion (EGP2). Whole-body insulin sensitivity was assessed with the euglycemic hyperinsulinemic clamp procedure; the use of 2 stepped insulin infusions and labeled glucose allowed the differentiation between hepatic and peripheral insulin sensitivity. EGP was measured under basal conditions; then during the low dose insulin infusion EGP was partially suppressed (hepatic insulin sensitivity), while during the high dose insulin infusion, EGP was almost completely suppressed and peripheral glucose uptake was maximally stimulated (peripheral insulin sensitivity).
Time Frame: 1 day
Population: All participants randomized and who had at least one euglycemic hyperinsulinemic clamp
Measure: Median (Full Range); unit: mg/kilogram (kg) body weight (BW)/min
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
mg/kilogram (kg) body weight (BW)/min
  Clamp 1 EGP0 | 1.79 [1.48 to 1.99]
  Clamp 1 EGP1 | 0.85 [0.51 to 0.98]
  Clamp 1 EGP2 | 0.07 [-0.02 to 0.36]
  Clamp 2 EGP0 | 1.68 [1.59 to 1.89]
  Clamp 2 EGP1 | 0.81 [0.71 to 0.98]

3. Primary Outcome: [6,6-2H2] Plasma Glucose Enrichment (PGE) in Part A
Description: [6,6-2H2] PGE was the molar fraction of labeled glucose measured in plasma. Whole-body insulin sensitivity was assessed with the euglycemic hyperinsulinemic clamp procedure; the use of 2 stepped insulin infusions and labeled glucose allowed the differentiation between hepatic and peripheral insulin sensitivity.
Time Frame: 1 day
Population: All participants randomized and who had at least one euglycemic hyperinsulinemic clamp
Measure: Mean (90% Confidence Interval); unit: percentage enrichment of plasma glucose
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
percentage enrichment of plasma glucose
  Clamp 1 | 2.96 [2.94 to 2.98]
  Clamp 2 | 2.97 [2.88 to 3.06]

4. Primary Outcome: Rate of Appearance of Glucose (Ra) in Part A
Description: Rate of appearance of glucose (Ra) in fasting state and during insulin infusions (Step 1 and Step 2).
Time Frame: 1 day
Population: All participants randomized and who had at least one euglycemic hyperinsulinemic clamp.
Measure: Mean (Full Range); unit: mg/kg BW/min
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
mg/kg BW/min
  Clamp 1 Step 1 | 3.575 [2.74 to 4.41]
  Clamp 1 Step 2 | 14.829 [9.90 to 19.76]
  Clamp 2 Step 1 | 2.859 [2.24 to 3.47]

5. Primary Outcome: Whole-body Glucose Uptake in Part A
Description: Whole-body glucose uptake (Rate of glucose disappearance, Rd) during the Step 2 Clamp
Time Frame: 1 day
Population: All participants randomized and who had at least one euglycemic hyperinsulinemic clamp.
Measure: Mean (90% Confidence Interval); unit: mg/kg BW/min
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
mg/kg BW/min | 14.829 [9.90 to 19.76]

6. Primary Outcome: Whole-body Glucose Uptake in Part B in Placebo Group
Description: Whole-body glucose uptake (Rate of glucose disappearance, Rd) during the Step 2 Clamp
Time Frame: 6 weeks
Population: Part B of the study was terminated due to the safety issue. Due to the limited participant number who completed study there no summary statistics were done by dosing regimen for Part B.
Measure: Mean (Full Range); unit: mg/kg BW/min
Arm/Group | Placebo - Part B
Number analyzed (Participants) | 6
mg/kg BW/min
  Step 2 Value 1 | 4.245 [4.18 to 4.41]
  Step 2 Value 2 | 6.325 [6.26 to 6.45]
  Step 2 Value 3 | 2.793 [2.72 to 2.85]
  Step 2 Value 4 | 6.835 [6.56 to 7.38]
  Step 2 Value 5 | 4.400 [3.97 to 5.23]
  Step 2 Value 6 | 3.940 [3.86 to 3.98]
  Step 2 Value 7 | 4.553 [4.37 to 4.62]
  Step 2 Value 8 | 4.225 [4.16 to 4.40]

7. Primary Outcome: Whole-body Glucose Uptake in Part B in PF-05175157 200 mg BID Group
Description: Whole-body glucose uptake (Rate of glucose disappearance, Rd) during the Step 2 Clamp
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: mg/kg BW/min
Arm/Group | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 7
mg/kg BW/min
  Step 2 Value 1 | 3.775 [3.70 to 3.83]
  Step 2 Value 2 | 9.033 [8.95 to 9.08]
  Step 2 Value 3 | 8.903 [8.33 to 9.37]
  Step 2 Value 4 | 11.310 [11.13 to 11.47]
  Step 2 Value 5 | 4.133 [3.98 to 4.50]
  Step 2 Value 6 | 6.763 [5.98 to 7.93]
  Step 2 Value 7 | 8.243 [8.06 to 8.73]
  Step 2 Value 8 | 7.180 [7.03 to 7.39]
  Step 2 Value 9 | 10.113 [9.80 to 10.28]
  Step 2 Value 10 | 6.205 [6.16 to 6.31]

8. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs), or Discontinuation Due to Adverse Events (AEs) in Part B
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline to follow-up (up to approximately 10 to 14 days after the last study drug administration)
Population: All participants who were admitted to the clinical research unit (CRU) on Day -5
Measure: Number; unit: Participants
Arm/Group | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 6 | 7
Participants
  Participants w ith AEs | 1 | 5
  Participants w ith SAEs | 0 | 1
  Participants discontinued due to AEs | 0 | 1

9. Primary Outcome: Number of Participants With Laboratory Test Abnormalities in Part B
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, and creatine phosphokinase); urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, and microscopy); others (follicle stimulating hormone [FSH], urine drug screen, lipid profile and very-low-density lipoproteins [VLDL], hemoglobin A1c [HbA1c], C-peptide, thyroid-stimulating hormone [TSH], Hepatitis B and C, human immunodeficiency virus [HIV], triglycerides, urine creatinine).
Time Frame: Screening up to follow-up (up to approximately 10 to 14 days after the last study drug administration)
Population: All participants who were admitted to the Clinical Research Unit (CRU) on Day -5
Measure: Number; unit: Participants
Arm/Group | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 6 | 7
Participants | 6 | 7

10. Primary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Categorical Summarization Criteria in Part B
Description: Criteria for potentially clinical important (PCI) change in vital signs included: sitting systolic blood pressure (SBP) of less than (<) 90 millimeters of mercury (mm Hg) or change in sitting SBP of greater or equal to (>=)30 mm Hg, sitting diastolic blood pressure (DBP) of <50 mm Hg or change in sitting DBP of >=20 mm Hg, sitting pulse rate of <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: Screening up to follow-up (up to approximately 10 to 14 days after the last study drug administration)
Population: All participants who were admitted to the CRU on Day -5
Measure: Number; unit: Participants
Arm/Group | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 6 | 7
Participants
  SBP <90 mm Hg | 0 | 0
  DBP <50 mm Hg | 0 | 0
  Pulse Rate <40 bpm | 0 | 0
  Pulse Rate >120 bpm | 0 | 0
  SBP maximum increase from baseline >=30 mm Hg | 0 | 0
  DBP maximum increase from baseline >=20 mm Hg | 0 | 0
  SBP maximum decrease from baseline >=30 mm Hg | 0 | 1
  DBP maximum decrease from baseline >=20 mm Hg | 0 | 0

11. Primary Outcome: Number of Participants With Change From Baseline and Absolute Values in Electrocardiogram (ECG) Meeting Categorical Summarisation Criteria in Part B
Description: Criteria for PCI changes in ECG (12-lead) were defined as: the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval) >=300 milliseconds (msec) and increase of >=25% from baseline when baseline >200 msec or increase of >=50% when baseline less than or equal to (<=) 200 msec; the time from the beginning of the electrocardiogram Q wave to the end of the S wave corresponding to ventricular depolarization (QRS interval) >=140 msec and increase of >=50% from baseline; the time corresponding to the beginning of depolarization to repolarization of the ventricles (QT), corrected for heart rate (QTc) using the Fridericia formula (QTcF) of 450 to < 480 msec and >=480 msec, or an increase from baseline of 30 to <60 msec or >=60 msec.
Time Frame: Screening up to follow-up (up to approximately 10 to 14 days after the last study drug administration)
Population: All participants who were admitted to the CRU on Day -5.
Measure: Number; unit: Participants
Arm/Group | Placebo - Part B | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 6 | 7
Participants
  QTc increase from Baseline of >=60 msec | 0 | 1
  QTcF increase from Baseline of >=60 msec | 0 | 1

12. Secondary Outcome: GIR in Part B in Placebo Group
Description: Glucose Infusion Rate rates obtained averaging respectively the last 30 minutes of glucose infusion at steady state on Step 1 (ie 150 to 180 min) and Step 2 (ie 330 to 360 min) insulin infusion.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: mg/min
Arm/Group | Placebo - Part B
Number analyzed (Participants) | 6
mg/min
  GIR1 Value 1 | 139.4 [0 to 150]
  GIR1 Value 2 | 178.3 [176 to 246]
  GIR1 Value 3 | 52.4 [0 to 97]
  GIR1 Value 4 | 196.5 [181 to 197]
  GIR1 Value 5 | 145.7 [92 to 161]
  GIR1 Value 6 | 104.7 [103 to 140]
  GIR1 Value 7 | 154.7 [143 to 218]
  GIR1 Value 8 | 85.4 [68 to 86]
  GIR2 Value 1 | 413.9 [411 to 461]
  GIR2 Value 2 | 645.0 [645 to 645]
  GIR2 Value 3 | 293.4 [217 to 296]
  GIR2 Value 4 | 668.2 [610 to 711]
  GIR2 Value 5 | 400.4 [368 to 504]
  GIR2 Value 6 | 359.3 [289 to 363]
  GIR2 Value 7 | 338.0 [338 to 338]
  GIR2 Value 8 | 343.3 [322 to 344]

13. Secondary Outcome: GIR in Part B in PF-05175157 200 mg BID Group
Description: as for outcome 12
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: mg/min
Arm/Group | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 7
mg/min
  GIR1 Value 1 | 170.5 [118 to 191]
  GIR1 Value 2 | 425.0 [367 to 427]
  GIR1 Value 3 | 334.2 [311 to 335]
  GIR1 Value 4 | 409.3 [277 to 521]
  GIR1 Value 5 | 50.0 [50 to 50]
  GIR1 Value 6 | 160.9 [160 to 188]
  GIR1 Value 7 | 113.2 [68 to 116]
  GIR1 Value 8 | 157.7 [113 to 225]
  GIR1 Value 9 | 215.2 [201 to 236]
  GIR1 Value 10 | 159.9 [159 to 178]
  GIR2 Value 1 | 359.2 [270 to 368]
  GIR2 Value 2 | 896.5 [871 to 921]
  GIR2 Value 3 | 896.3 [864 to 1064]
  GIR2 Value 4 | 1078.5 [1068 to 1079]
  GIR2 Value 5 | 357.6 [357 to 370]
  GIR2 Value 6 | 564.0 [520 to 656]
  GIR2 Value 7 | 693.1 [666 to 728]
  GIR2 Value 8 | 647.2 [623 to 681]
  GIR2 Value 9 | 889.4 [821 to 893]
  GIR2 Value 10 | 519.5 [512 to 540]

14. Secondary Outcome: EGP in Part B in Placebo Group
Description: EGP measured by means of euglycemic hyperinsulinemic clamp preceding insulin infusion (EGP0), on Step 1 insulin infusion (EGP1) and on Step 2 insulin infusion (EGP2)
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/kg fat free mass (FFM)/min
Arm/Group | Placebo - Part B
Number analyzed (Participants) | 6
mg/kg fat free mass (FFM)/min
  EGP0 Value 1 | 1.540 [1.49 to 1.60]
  EGP0 Value 2 | 1.690 [1.64 to 1.75]
  EGP0 Value 3 | 1.285 [1.24 to 1.33]
  EGP0 Value 4 | 1.575 [1.55 to 1.62]
  EGP0 Value 5 | 1.965 [1.89 to 2.04]
  EGP0 Value 6 | 1.538 [1.50 to 1.58]
  EGP0 Value 7 | 1.518 [1.47 to 1.56]
  EGP0 Value 8 | 1.518 [1.49 to 1.56]
  EGP1 Value 1 | 0.600 [0.57 to 0.66]
  EGP1 Value 2 | 0.585 [0.55 to 0.61]
  EGP1 Value 3 | 0.525 [0.49 to 0.59]
  EGP1 Value 4 | 0.500 [0.49 to 0.52]
  EGP1 Value 5 | 0.808 [0.75 to 0.86]
  EGP1 Value 6 | 0.830 [0.82 to 0.84]
  EGP1 Value 7 | 0.560 [0.55 to 0.58]
  EGP1 Value 8 | 0.825 [0.78 to 0.85]
  EGP2 Value 1 | 0.200 [0.17 to 0.22]
  EGP2 Value 2 | -0.063 [-0.09 to -0.03]
  EGP2 Value 3 | -0.050 [-0.10 to -0.01]
  EGP2 Value 4 | 0.280 [0.25 to 0.31]
  EGP2 Value 5 | 0.145 [0.06 to 0.23]
  EGP2 Value 6 | 0.223 [0.20 to 0.24]
  EGP2 Value 7 | 0.180 [0.17 to 0.19]
  EGP2 Value 8 | 0.405 [0.38 to 0.46]

15. Secondary Outcome: EGP in Part B in PF-05175157 200 mg BID Group
Description: as for outcome 14
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/kg fat free mass (FFM)/min
Arm/Group | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 7
mg/kg fat free mass (FFM)/min
  EGP0 Value 1 | 1.240 [1.23 to 1.27]
  EGP0 Value 2 | 1.445 [1.42 to 1.46]
  EGP0 Value 3 | 2.083 [2.03 to 2.15]
  EGP0 Value 4 | 1.708 [1.68 to 1.73]
  EGP0 Value 5 | 1.695 [1.67 to 1.72]
  EGP0 Value 6 | 1.615 [1.59 to 1.65]
  EGP0 Value 7 | 1.690 [1.64 to 1.75]
  EGP0 Value 8 | 1.393 [1.25 to 1.46]
  EGP0 Value 9 | 1.448 [1.43 to 1.46]
  EGP0 Value 10 | 1.345 [1.33 to 1.36]
  EGP1 Value 1 | 0.568 [0.54 to 0.59]
  EGP1 Value 2 | 0.250 [0.22 to 0.28]
  EGP1 Value 3 | 0.788 [0.69 to 0.89]
  EGP1 Value 4 | 0.575 [0.54 to 0.62]
  EGP1 Value 5 | 1.183 [1.12 to 1.22]
  EGP1 Value 6 | 0.538 [0.52 to 0.55]
  EGP1 Value 7 | 0.765 [0.74 to 0.78]
  EGP1 Value 8 | 0.555 [0.53 to 0.58]
  EGP1 Value 9 | 0.193 [0.11 to 0.23]
  EGP1 Value 10 | 0.418 [0.35 to 0.45]
  EGP2 Value 1 | 0.253 [0.23 to 0.29]
  EGP2 Value 2 | 0.165 [0.09 to 0.21]
  EGP2 Value 3 | -0.035 [-0.43 to 0.14]
  EGP2 Value 4 | 0.243 [0.10 to 0.39]
  EGP2 Value 5 | 0.543 [0.47 to 0.67]
  EGP2 Value 6 | 0.110 [0.03 to 0.15]
  EGP2 Value 7 | 0.190 [0.15 to 0.24]
  EGP2 Value 8 | -0.313 [-0.42 to -0.23]
  EGP2 Value 9 | -0.253 [-0.34 to -0.20]
  EGP2 Value 10 | 0.198 [0.19 to 0.21]

16. Secondary Outcome: Ra in Part B in Placebo Group
Description: Ra in fasting state and during insulin infusions (Step 1 and Step 2).
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: mg/kg BW/min
Arm/Group | Placebo - Part B
Number analyzed (Participants) | 6
mg/kg BW/min
  Step 2 Value 1 | 4.245 [4.18 to 4.41]
  Step 2 Value 2 | 6.325 [6.26 to 6.45]
  Step 2 Value 3 | 2.793 [2.72 to 2.85]
  Step 2 Value 4 | 6.835 [6.56 to 7.38]
  Step 2 Value 5 | 4.400 [3.97 to 5.23]
  Step 2 Value 6 | 3.940 [3.86 to 3.98]
  Step 2 Value 7 | 4.553 [4.37 to 4.62]
  Step 2 Value 8 | 4.225 [4.16 to 4.40]

17. Secondary Outcome: Ra in Part B in PF-05175157 200 mg BID Group
Description: Ra in fasting state and during insulin infusions (Step 1 and Step 2).
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: mg/kg BW/min
Arm/Group | PF-05175157 200 mg Twice a Day - Part B
Number analyzed (Participants) | 7
mg/kg BW/min
  Step 2 Value 1 | 3.775 [3.70 to 3.83]
  Step 2 Value 2 | 9.033 [8.95 to 9.08]
  Step 2 Value 3 | 8.903 [8.33 to 9.37]
  Step 2 Value 4 | 11.310 [11.13 to 11.47]
  Step 2 Value 5 | 4.133 [3.98 to 4.50]
  Step 2 Value 6 | 6.763 [5.98 to 7.93]
  Step 2 Value 7 | 8.243 [8.06 to 8.73]
  Step 2 Value 8 | 7.180 [7.03 to 7.39]
  Step 2 Value 9 | 10.113 [9.80 to 10.28]
  Step 2 Value 10 | 6.205 [6.16 to 6.31]

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (up to approximately 3 days after the last clamp procedure in Part A and up to approximately 10 to 14 days after the last study drug administration in Part B)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | All Participants in Part A | PF-05175157 200 mg Twice a Day - Part B | Placebo - Part B
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 5/7 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants in Part A (N=6) | PF-05175157 200 mg Twice a Day - Part B (N=7) | Placebo - Part B (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants in Part A (N=6) | PF-05175157 200 mg Twice a Day - Part B (N=7) | Placebo - Part B (N=6)
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Part B of the study was terminated due to the safety issue. Due to the low number of participants who completed the study, there are no conclusions for PK or PD in Part B. The prioritization of Part A endpoints was done by inputs from team.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.